CLINICAL TRIAL: NCT04095663
Title: Comparison of Surgery and Medicine on the Impact of Diverticulitis (COSMID) Trial
Acronym: COSMID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, David Flum, Professor, School of Medicine: Surgery, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007409
Record Dates: First submitted 2019-08-28; First posted 2019-09-19 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Diverticulitis
MeSH Terms: conditions — Diverticulitis | interventions — Practice Management, Medical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partial Colectomy (Active Comparator): Elective segmental colectomy for diverticular disease involves removal of the segment of colon (most commonly sigmoid and/or left colon) where there has been disease identified by computed tomography imaging or colonoscopy. Elective colectomy usually removes the affected colon along with adjacent segments that have diverticula, with a primary anastomosis performed to reestablish bowel continuity. Most surgeons now perform the procedure using a laparoscopic approach, when possible, and sometimes use a temporary, protective stoma if the re-connection is considered high-risk. The technique for laparoscopic resection is not specified by the protocol (allows for any number of laparoscopic port sites, all incision types, hand-assistance and robotic) with details of the technique recorded. If randomized to elective colectomy, patients will be encouraged to undergo the procedure within 6 weeks of assignment.
  Interventions: Procedure: Partial Colectomy
- Medical Management (Active Comparator): Medical management for diverticular disease has been used for over 30 years and includes a set of interventions, all components of which have been the subject of small, but often positive trials. All patients randomized to medical management or who select it as their treatment in the observational cohort will view a video (provided in English and Spanish) that explains each element of the medical management "toolbox": diet and exercise recommendations, fiber supplementation (e.g., augmenting dietary fiber or over the counter fiber supplements), with mesalazine tablets or suppositories, probiotics and rifamycin. In consultation with their physician, they will be recommended to a regimen of diet and exercise and fiber supplementation. Clinicians will be asked to consider rifamycin (dose/frequency) for those with AUD who are not responding to diet and exercise and mesalazine (dose/frequency) for those with lingering symptoms who are not responding to diet and exercise.
  Interventions: Other: Medical Management

INTERVENTIONS:
Procedure: Partial Colectomy — Most partial colectomies are performed using a laparoscopic approach, when possible, and surgeons sometimes use a temporary, protective stoma if the re-connection is considered high risk.
  Arms: Partial Colectomy
Other: Medical Management — Patients will be offered a varying combination of tools from the best medical management "toolbox" (diet and exercise, fiber supplementation/probiotics, and rifamycin/mesalazine) depending on what they have already tried. Based on the "evidence-based best medical toolbox" clinicians will be asked to consider rifamycin (dose/frequency) for those with AUD who are not responding to diet and exercise and mesalazine (dose/frequency) for those with lingering symptoms who are not responding to diet and exercise.
  Arms: Medical Management

SUMMARY:
The COSMID (Comparison of Surgery and Medicine on the Impact of Diverticulitis) trial is a pragmatic, patient-level randomized superiority trial of elective colectomy vs. best medical management for patients with quality of life (QoL) limiting diverticular disease. A parallel observational cohort will include those who are disinclined to have their treatment choice randomized, but are willing to contribute information about their outcomes. The goal of the COSMID trial is to answer the question: For patients with QoL-limiting diverticular disease, is elective colectomy more effective than best medical management? The hypothesis being tested in the COSMID trial is that patient-reported outcomes (PROs) among patients in the surgery arm will be superior to those in the best medical management arm.

DETAILED DESCRIPTION:
For over 50 years, professional society recommendations for the management of uncomplicated diverticulitis included early elective surgery to prevent the need for an emergency operation and avoid the risk of colostomy. Over the last 15 years the notion that a patient must have a certain number of episodes of acute uncomplicated diverticulitis (AUD) before undergoing elective colectomy has changed dramatically. This was, in part, due to studies showing that emergency surgery for complicated disease is much more likely to be needed during the first episode of diverticulitis, making the notion of prophylactic elective colectomy for AUD less relevant. Furthermore, clinicians realized that most recurrent episodes of AUD could be managed with outpatient antibiotics alone and that "best medical management" - including fiber supplementation, mesalazine, rifamycin and probiotics - could reduce symptoms between episodes of AUD. All of the components of best medical management have some, albeit limited, evidence of effectiveness, most in improving symptoms rather than reducing the risk of recurrence and are relatively safe and inexpensive. Best medical management is far less invasive than elective surgery but infrequently prescribed the US, in part because of limited insurance coverage. Alternatively, resection removes the diseased segment of colon, does relieve symptoms and decreases the risk of recurrence.

In 2014, guidelines from the American Society of Colorectal Surgeons (ASCRS) abandoned "episode count" as an indication for surgery in patients with AUD and instead recommended individualizing the decision to operate for AUD based on the "effects on lifestyle (professional and personal) of recurrent attacks". Decision making about surgery in patients with lingering symptoms after recovery from an episode of AUD has not been the specific focus of an ASCRS guideline, but recommendations about elective surgery emphasize individualizing decision making based on the overall impact of the disease on the patient.These recommendations for individualization of treatment based on the quality of life (QoL) impact of recurrent AUD and lingering symptoms highlight the decision that hundreds of thousands of people now have to make each year. Based on the effect of the disease on their QoL they must choose between two very different treatment options: elective colectomy vs. best medical management. While the recommendation to individualize treatment based on the QoL impact is a step forward in advancing patient-centered care, the comparative effectiveness of these two treatments on symptoms and QoL has not been well studied.

This will be a multi-site, open randomized trial in which participants with either recurrent AUD or lingering symptoms after an episode of AUD are randomized to one of two initial treatment strategies, elective segmental colectomy (performed laparoscopically when possible) and best medical management.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years
* At least one episode of diverticulitis confirmed by CT scan and a colonoscopy (completed or scheduled) to rule out or screen for other colon pathology in accordance with colorectal cancer screening guidelines
* Persistent signs, symptoms, or concerns related to diverticulitis after recovery from an episode of left-sided diverticulitis
* Self-reported QoL limitation (assessed with 12 questions modified from the Diverticulitis Quality of Life [DV-QOL] instrument).

Exclusion Criteria:

* Unable to consent in English or Spanish
* Current diagnosis or previous endoscopic or surgical interventions for fistula, or stricture or current significant bleeding, related to diverticulitis
* Last episode of acute diverticulitis currently unresolved (i.e., on antibiotics for diverticulitis; drain in place)
* Previous operation for diverticulitis
* Right-sided diverticulitis
* Immunodeficiency (e.g., absolute neutrophil count <500/mm3, chronic immunosuppressive drugs like oral corticosteroids, anti-TNF agents, or known AIDS [i.e., recent CD4 count <200] assessed by patient history)
* Actively undergoing chemotherapy or radiation for malignancy
* Expectant or concurrent hemodialysis, peritoneal dialysis, treatments using indwelling venous catheters, or conditions putting patient at risk for bacterial seeding
* Diagnosis of inflammatory bowel disease (i.e., Crohn's, ulcerative colitis)
* Taking prescription medication for irritable bowel syndrome
* Intolerance or allergy to all medications in the medical management arm
* Surgeon is unwilling to offer surgery due to comorbid or prior surgical conditions that contraindicate elective surgery (e.g., liver failure, renal failure, malignancy, "frozen abdomen")
* Abdominal/pelvic surgery within the past month
* Pregnant or expecting to become pregnant in the 30 days following baseline/screening
* Unable to consent to research or self-respond to follow-up surveys (e.g., altered mental status)
* Currently incarcerated in a detention facility or in police custody at baseline/screening (patients wearing a monitoring device can be enrolled)
* Prior enrollment in the COSMID study or planning on enrollment in another investigational drug or vaccine while on study treatment
* Unable or unwilling to return, be contacted for, or complete research surveys.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Patient-reported quality of life as measured by Gastrointestinal Quality of Life Index (GIQLI) | Mean GIQLI at 6, 9, and 12 months following randomization to treatment
  A 36-item questionnaire assessing 5 domains: GI symptoms, physical function, emotional well-being, social well-being, and perception of medical treatment measured by a single item question. Each item has 5 response choices (i.e., all of the time, most of the time, some of the time, a little of the time, never). In addition, the measure produces an overall quality of life score (0-144) where higher numbers indicate greater QoL.

SECONDARY OUTCOMES:
Diverticulitis Quality of Life (DV-QoL) instrument | Baseline, 12 months, 24 months
  A 17-item questionnaire including a pain scale and questions about about physical, emotional, and social effects of diverticulitis over the past 2 weeks, with a total score ranging from 0 (best) to 10 (worst) with higher scores reflecting worse quality of life effects from diverticulitis.
Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health measure | Baseline; 6, 12, 24, 36 months
  A 10-item instrument measuring domains that can be scored into a Global Physical Health component and Global Mental Health component. Each item includes 5 response choices, with the exception of the common 11-point pain intensity item ("How would you rate your pain on average?" with 0=no pain and 10=worst imaginable pain), where higher scores reflect more severe symptoms/impairment.
Decision Regret Scale | 6 and 36 months
  A 5-item validated questionnaire that measures regret among patients following a specific treatment decision. Scores range from 0-100 and higher scores reflect higher levels of regret. While developed for use in patients undergoing treatment for cancer, the questions are general in nature and adaptable to diverse clinical experiences.
Work Productivity and Activity Impairment instrument | Baseline; 6, 12, 18, 24, 30, 36 months
  A 6-item instrument used to measure the effect of general health and symptom severity on work productivity and regular activities during the past seven days. Scores are calculated applying algorithms to the five numerical responses, three of which are continuous variables (hours) and two of which are a scale from 0-10, then converting to a percentage, with higher WPAI scores indicating greater impairment and less productivity.
  The WPAI measures work productivity loss due to general health or a specified health problem. This questionnaire has been validated for use in many gastrointestinal diseases, including gastroesophageal reflux disease, irritable bowel syndrome, and Crohn's disease.

CONTACTS AND LOCATIONS:
Overall Officials: David R Flum, MD, Principal Investigator — University of Washington
Locations (29):
- United States (29):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UC San Diego Health, San Diego, California
  - UCSF Health, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Memorial Health University Medical Center, Savannah, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Northwestern University, Evanston, Illinois
  - University of Iowa Healthcare, Iowa City, Iowa
  - Boston University Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Albany Medical College, Albany, New York
  - New York Presbyterian-Queens, Flushing, New York
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Atrium Health-Carolinas Medical Center, Charlotte, North Carolina
  - Mount Carmel Health Systems, Columbus, Ohio
  - Penn Medicine, Philadelphia, Pennsylvania
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - UTHealth Houston, Houston, Texas
  - University of Utah Health, Salt Lake City, Utah
  - VCU Medical Center, Richmond, Virginia
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data and results from this proposal stand to develop research that may have a lasting value beyond the term of the award and will be archived and preserved, supporting access to third parties interested in replication and verification of our results and data reuse by other investigators planning future studies. We will prepare and share a complete, cleaned, de-identified copy of the final dataset used in conducting the final analyses upon which the accepted primary study publication is based. The final dataset will include participants' treatment group assignment, demographics and patient reported outcomes (GIQLI survey). Data collected on clinical variables will also include: NSQIP-defined complications major complications, dates and details of healthcare utilization including hospitalizations, length of stay, use of imaging, colectomy details and associated pathology results, and medication use.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: We intend to prepare and share a complete, cleaned, de-identified copy of the final dataset used in conducting the final analyses upon which the accepted primary study publication is based, timing dependent on funding. Our goal is that data will be made available no later than the end of the completion of the funded project period for the parent award or once a manuscript (or manuscripts) covering the primary study aims have been published, whichever is earlier. A complete study data set will be permanently archived and available through the PCODR as described above.
Access Criteria: Aggregate clinical trials data from all arms of the study will be available in ClinicalTrials.gov, along with related metadata. All other data described above in the "data to be shared" section will be available through the PCODR and preserved through methods which are in accordance with standard practice. There are no anticipated factors or limitations that will affect the access, distribution or reuse of the scientific data generated by the proposal. Data will be shared as allowed by the participant's informed consents and in accord with IRB approval.

REFERENCES:
- [Derived] Hantouli MN, Schmicker RH, Tufte JE, Ali FG, Bennett RD, Cohan JN, Comstock BA, Curran T, Davidson GH, Eisenstein S, Fischkoff KN, Fleming FJ, Gribovskaja-Rupp I, Jafari MD, Kessler LG, Krane MK, Lawrence SO, McCormick JT, Millas SG, Morris AM, Pullar KM, Reinke CE, Saraidaridis JT, Simianu VV, Watkins SP, White NB, Wick EC, Wieghard N, Flum DR, Read TE; COSMID Collaborative. Comparison of Surgery and Medicine on the Impact of Diverticulitis (COSMID) trial: a protocol for a pragmatic randomised study of diverticulitis treatment in the USA. BMJ Open. 2026 Jan 8;16(1):e098309. doi: 10.1136/bmjopen-2024-098309. PMID 41506759